CLINICAL TRIAL: NCT03678948
Title: Evaluation of the Efficacy of Radiofrequency-Based Debridement vs. Mechanical Debridement for the Treatment of Articular Cartilage Lesions
Brief Title: Radiofrequency-Based Debridement vs. Mechanical Debridement for the Treatment of Articular Cartilage Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discontinuing research
Sponsor: Christopher Kaeding (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christopher Kaeding, Professor - Clinical, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018H0244
Record Dates: First submitted 2018-08-30; First posted 2018-09-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Articular Cartilage Disorder of Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study subject will not be made aware of the treatment received until after completion of the research study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Radiofrequency-Based Debridement (Active Comparator): The Smith and Nephew WEREWOLF COBLATION System is indicated for all soft tissue types in the knee. The WEREWOLF COBLATION System is a FDA cleared bipolar, radiofrequency electrosurgical system designed for use in orthopaedic/arthroscopic surgical procedures.
  Interventions: Device: Radiofrequency-Based Debridement
- Mechanical Debridement (Active Comparator)
  Interventions: Device: Mechanical Debridement

INTERVENTIONS:
Device: Radiofrequency-Based Debridement — In this process, radiofrequency energy is used to excite the water molecules in a conductive medium, such as an electrolyte (saline) solution, to generate excited radicals within precisely focused plasma. The energized particles in the plasma have sufficient energy to break molecular bonds (16-18), excising or dissolving (i.e. ablating) soft tissue at relatively low temperatures (typically 40ºC to 70ºC).
  Other Names: Werewolf Coblation Wand
  Arms: Radiofrequency-Based Debridement
Device: Mechanical Debridement — Arthroscopic chondroplasty used to remove loose and damaged cartilage which minimizes synovial irritation and mechanical impingement
  Arms: Mechanical Debridement

SUMMARY:
The purpose of this study is to evaluate the changes in clinical and imaging outcomes following arthroscopic treatment of chondral lesion(s) by Radiofrequency-Based debridement or Mechanical Debridement in subjects 18-50 years of age.

DETAILED DESCRIPTION:
This is a non-inferiority, prospective, single blinded, randomized, single-center study design with enrollment of 82 randomized subjects (to assure 70 subjects complete the study). The sample size of 82 participants was calculated from a power analysis. The study was powered to detect at least a seven point change in KOOS pain score based on achieving 80% statistical power to detect a non-inferiority margin. Study duration will be until the last subject enrolled reaches 52 weeks post-operative.

The 82 randomized subjects will be randomized at a 1:1 ratio into the Werewolf Coblation wand treatment group or mechanical debridement treatment group. Subjects will be blinded to their treatment assignment until they complete all study visits. Upon withdraw from the study, termination from the study, or new or recurrent symptoms requiring a subsequent arthroscopy, the blinded assignment will be revealed to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent on the IRB approved consent form specific to the study, prior to study participation
* 18-50 years old
* Male or Female
* Suspected chondral damage in the following locations where debridement is indicated:

  * Medial femoral condyle
  * Lateral femoral condyle
  * Trochlea
  * Patella
* < 30% joint space narrowing as seen on x-ray (merchant view, AP and PA Rosenberg)
* 1 or more chondral lesion(s) as noted on MRI

Exclusion Criteria:

* Previous chondral treatment in the same compartment (prior debridement and lavage performed more than three months prior to baseline are acceptable)
* Focal chondral defect indicated for concomitant procedures (i.e., microfracture, ACI, MACI, OATs)
* Concomitant procedures that are not allowed:

  * Lateral retinacular release
  * Excision of osteophytes
  * Subchondroplasty
  * Manipulation under anesthesia
  * ACL reconstruction
  * Quad tendon repair
  * Patellar tendon repair
  * Patellar tendon debridement
  * Multiligament reconstruction
* Pregnant and/or intending to become pregnant during this study period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Knee and Osteoarthritis Outcome Scores (KOOS) activity subscale | change from baseline at week 52 post-op
  The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | change from baseline at week 52 post-op
  Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
International Knee Documentation Committee (IKDC) subjective knee evaluation | change from baseline at week 52 post-op
International Knee Documentation Committee (IKDC) objective knee | change from baseline at week 52 post-op
Marx Activity Rating Scale (MARS) | change from baseline at week 52 post-op
  MARS includes 4 items that assess the frequency of running, cutting, decelerating, and pivoting based on the subjects "healthiest and most active state in the past year." A higher score indicates more functional demand on the knee joint and potentially a higher risk of injury. Each item is scored on a 5-point ordinal scale ranging from 0 (less than 1 time in a month) to 4 (4 or more times in a week), and the total scale score is obtained by summing the individual items' scores (range, 0-16).
Work Productivity and Activity Impairment (WPAI V2.0) | change from 1 week post op to 6 weeks post-op
  Asks about the effect of patient knee injury on their ability to work and perform normal daily activities
MRI | change from baseline at week 52 post-op
  Baseline MRI will be compared to MRI at 52 weeks to evaluate knee morphology, cartilage signal, osteophytes, bone marrow edema, subarticular cysts, effusions and loose bodies. The international cartilage repair score will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kaeding, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center Jameson Crane Sports Medicine Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT03678948/Prot_001.pdf
  • Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT03678948/ICF_000.pdf